CLINICAL TRIAL: NCT00025376
Title: A Phase II Trial of PS-341 in Patients With Renal Cell Cancer
Brief Title: PS-341 in Treating Patients With Metastatic Kidney Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11049A; UCCRC-11049A; NCI-3291
Record Dates: First submitted 2001-10-11; First posted 2003-06-17 (Estimated); Last update posted 2013-09-05 (Estimated); Status verified 2013-09

CONDITIONS: Kidney Cancer
Keywords: stage IV renal cell cancer; recurrent renal cell cancer
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell | interventions — Bortezomib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Pre-Treatment biopsy followed by PS-341 administration (Experimental): Pre-treatment tumor biopsy followed by 3 cycles of PS-341 given by IV infusion. Each cycle will last 3 weeks. PS-341 will be given 2 times a week for 2 weeks followed by a 'rest' week with no drug. After the 3rd cycle, subjects can continue to receive another 3 cycles of the study drug if their disease has not worsened.
  Interventions: Drug: PS-341; Procedure: Tumor Biopsy
- PS-341 administration followed by biopsy (Experimental): 3 cycles of PS-341 given by IV infusion. Each cycle will last 3 weeks. PS-341 will be given 2 times a week for 2 weeks followed by a 'rest' week with no drug. After the 3rd cycle, subjects will have a tumor biopsy and can continue to receive another 3 cycles of the study drug if their disease has not worsened.
  Interventions: Drug: PS-341; Procedure: Tumor Biopsy

INTERVENTIONS:
Drug: PS-341
Procedure: Tumor Biopsy

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. It is not yet known which regimen of PS-341 is more effective in treating metastatic kidney cancer.

PURPOSE: Randomized phase III trial to study the effectiveness of PS-341 in treating patients who have metastatic kidney cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the objective response rate in patients with metastatic renal cell cancer treated with bortezomib.
* Determine the time to tumor progression and 1-year survival of patients treated with this drug.
* Determine the toxicity profile of this drug in these patients.

OUTLINE: This is a randomized, multicenter study. Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive bortezomib IV over 3-5 seconds twice weekly on weeks 1 and 2. Treatment repeats every 3 weeks for 3 courses in the absence of disease progression or unacceptable toxicity. Patients then undergo core biopsy.
* Arm II: Patients undergo core biopsy. Patients then receive bortezomib IV as in arm I.

Patients undergo radiologic re-evaluation of measurable lesions. Patients with stable disease or a partial or complete response continue to receive bortezomib in the absence of disease progression or unacceptable toxicity.

Patients are followed for 2 years.

PROJECTED ACCRUAL: A total of 21-41 patients will be accrued for this study within 9-14 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed metastatic renal cell cancer
* Measurable disease

  * At least 2.0 cm in at least 1 dimension by physical exam OR at least 1.0 cm in at least 1 dimension by radiologic exam
  * Single measurable lesion must not be within prior radiotherapy portal
* Tumor lesion amenable to core biopsy

  * At least 1 cm of tumor obtainable
* No active CNS metastatic disease

  * Single previously resected CNS metastasis allowed provided no disease progression 8 weeks after therapy and no longer requiring steroids or antiseizure medications

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* Not specified

Life expectancy:

* More than 3 months

Hematopoietic:

* WBC at least 3,000/mm^3
* Absolute neutrophil count at least 1,500/mm^3
* Platelet count at least 100,000/mm^3

Hepatic:

* Bilirubin no greater than 1.5 times upper limit of normal (ULN)
* AST/ALT no greater than 2.5 times ULN

Renal:

* Creatinine no greater than 2.0 mg/dL

Cardiovascular:

* No symptomatic congestive heart failure
* No unstable angina pectoris
* No cardiac arrhythmia

Other:

* No other uncontrolled concurrent illness
* No ongoing or active infection
* No psychiatric illness or social situation that would preclude study compliance
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective barrier-method contraception during and for 3 months after study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Prior immunotherapy or biotherapy allowed

Chemotherapy:

* No prior chemotherapy

Endocrine therapy:

* See Disease Characteristics

Radiotherapy:

* See Disease Characteristics
* At least 4 weeks since prior radiotherapy
* No prior radiotherapy to 25% or more of bone marrow (i.e., whole pelvis)

Surgery:

* See Disease Characteristics

Other:

* No other concurrent investigational agents
* No concurrent combination antiretroviral therapy for HIV-positive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2001-10; Primary Completion 2002-09 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Response Rate of PS-341 in colon cancer | 9 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Walter M. Stadler, MD, FACP, Study Chair — University of Chicago
Locations (10):
- United States (10):
  - University of Chicago Cancer Research Center, Chicago, Illinois
  - Louis A. Weiss Memorial Hospital, Chicago, Illinois
  - Cancer Care Specialists of Central Illinois, S.C., Decatur, Illinois
  - Ingalls Memorial Hospital, Harvey, Illinois
  - LaGrange Memorial Hospital, LaGrange, Illinois
  - Loyola University Medical Center, Maywood, Illinois
  - Oncology/Hematology Associates of Central Illinois, P.C., Peoria, Illinois
  - Fort Wayne Medical Oncology and Hematology, Inc., Fort Wayne, Indiana
  - Michiana Hematology/Oncology P.C., South Bend, Indiana
  - Oncology Care Associates, P.L.L.C., Saint Joseph, Michigan